CLINICAL TRIAL: NCT01230788
Title: A Trial of Rituximab Combined With Prednisone/Ifosfamide/Etoposide for Relapsed Acute Lymphoblastic Leukemia (ALL)
Brief Title: Rituximab for Patients With Relapsed Acute Lymphoblastic Leukemia
Acronym: Rituximab
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Todd M. Cooper, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00039682; Rituximab (Other: Other)
Record Dates: First submitted 2010-10-23; First posted 2010-10-29 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Leukemia; Acute Lymphoblastic Leukemia; ALL
Keywords: ALL; Leukemia; Rituximab; Pediatrics
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab (Experimental): study drug given
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — 375 mg/m2/dose on days 8, 15, 22, and 29 (diluted in NS to a final concentration of 1 mg/ml for ease of administration). (Premedicate with Acetaminophen 15 mg/kg po (max 650 mg) and Diphenhydramine 1 mg/kg IV/PO (max 50 mg)).

SUMMARY:
This is a pilot study of a drug called rituximab used together with other drugs-prednisone, etoposide, and ifosfamide. Prednisone, etoposide, and ifosfamide have been used as part of standard chemotherapy for relapsed Acute Lymphoblastic Leukemia (ALL). Rituximab was approved by the Food and Drug Administration in 1997. However, the use of rituximab with prednisone, etoposide, and ifosfamide in pediatric patients with relapsed or refractory ALL is considered experimental.

This study is for patients who have ALL in second or greater relapse, or in first relapse and not responding to treatment.

The goals of this study are:

* To see if using rituximab with prednisone, etoposide, and ifosfamide is beneficial to leukemia treatment
* To find out what side effects this combination of drugs can cause

A total of 15 participants (30 years old or younger) will be enrolled, over a period of 2 years.

DETAILED DESCRIPTION:
Rationale for study design:

The combination of etoposide and ifosfamide is a reinduction regimen used in many previous studies for pediatric B lineage acute lymphoblastic leukemia (ALL). It does not use anthracyclines, and therefore can be safely used in patients at risk for cardiac toxicity due to previous anthracycline use.

Previous studies in adult patients with ALL have demonstrated safety and efficacy with the addition of rituximab to other induction regimens. Rituximab is an anti-CD20 monoclonal antibody. Approximately one-half of pediatric cases of B precursor ALL express the CD20 antigen on the leukemic blasts. The use of rituximab provides a potential target for CD20 positive cells, therefore improving the rates of cytotoxicity associated with the chemotherapy. Rituximab has been previously utilized in many pediatric and adult regimens in combination with other chemotherapeutic agents, and is expected to be safe with the combination of etoposide and ifosfamide. However, since it has never been studied with this combination of chemotherapy, strict stopping rules are in place to ensure that it is a safe combination.

A recent study demonstrated upregulation of CD20 expression on leukemic blasts exposed to one week of prednisone therapy. This increase in expression occurred in the majority of B-ALL patient samples, regardless of whether the patient initially expressed CD20 on the surface of the leukemic blasts. In those samples with upregulation of CD20 treated with rituximab, cytotoxicity from rituximab was more successful than in samples with a smaller percentage of CD20 expression.

Therefore, prednisone will be given for two weeks in combination with etoposide and ifosfamide. It is hoped that the percentage of leukemic blasts expressing CD20 will increase with this combination of medications, allowing the rituximab to be more effective when given weekly starting on day 8 of therapy. To better understand this process, samples of blood and bone marrow will be collected to quantify CD20 expression and the amount of leukemia present at multiple time points during the month of study duration.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients must be 1-30 years of age at initial diagnosis.
2. Diagnosis: Patients must have histologically-confirmed relapsed/refractory Acute Lymphoblastic Leukemia (ALL).
3. Disease Status:Patients must be in

   * second or greater bone marrow relapse (≥ 25% blasts by morphology), or
   * refractory to reinduction therapy with one or more attempts at remission reinduction (end of reinduction blasts ≥ 5% by morphology and/or end of reinduction MRD ≥ 1% by flow cytometry).
   * Patients with combined bone marrow and extramedullary relapse are eligible (CNS 3 patients excluded).
4. Performance Status: Patients must have a performance status of ≥50 from the Lansky Scale if <10 years or ≥ 50 or from the Karnofsky Scale if ≥ 10 years. Patients who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.
5. Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study and meet time restrictions from end of prior therapy as stated below:

   * Myelosuppressive chemotherapy: must not have received within 2 weeks of entry onto this study (4 weeks in the case of nitrosurea containing therapy). Patients who relapse while receiving ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study. Cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of therapy.
   * XRT: must be ≥ 4 weeks since the completion of radiation therapy.
   * Study specific limitations: must be ≥ 7 days since the completion of corticosteroid therapy.
   * Growth factor(s): Must not have received any hematopoietic growth factors (GCSF, Neulasta, or GMCSF) within 7 days of study entry.
   * Stem Cell Transplant: Patients must be at least two months from stem cell transplant, must be off immunosuppressives, and must have no evidence of active graft versus host disease.

   Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
6. Institutional review board approval.
7. Individual informed consent per local guidelines and federal and state regulations.
8. Organ Function: All patients must have adequate organ function defined as:

   * Renal Function: Patients must have a calculated creatinine clearance or radioisotope GFR ≥ 70mL/min/1.73m2 or a normal serum creatinine based on age/gender.
   * Liver Function: Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) for age, AND SGPT (ALT) ≤ 5 x institutional ULN for age
   * Cardiac Function: Ejection fraction > 50% on echocardiogram or MUGA Scan, OR Shortening fraction ≥ 27% on echocardiogram or MUGA Scan
   * Reproductive Function: Due to potential teratogenic effects of the drugs, all post-menarchal female patients must have a negative serum beta HCG prior to study enrollment. In addition, all patients of childbearing or child-fathering potential must agree to a medically acceptable form of contraception, including abstinence, while on study.

Exclusion Criteria:

1. Patients with an active and uncontrolled infection, defined as need for pressors, and/or positive cultures for 24 hours.
2. Patients recovering from allogeneic bone marrow transplantation who are still on immunosupressants.
3. Pregnant or lactating females. Women of childbearing age will agree to use contraception during the protocol.
4. Patients currently receiving other investigational agents, medications, or supplements with a known anti-leukemic effect.
5. Patients who, in the opinion of the investigator, will not be able to comply with safety monitoring requirements of the study.
6. Patients with reactivation of hepatitis B prior to starting therapy.
7. Patients who are HIV positive.
8. Patients must not have CNS 3 involvement.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Cooper, DO, Principal Investigator — Emory University/Children's Healthcare of Atlanta
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - The children's Mercy Hospital, Kansas City, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant recruited between September 2010 and June 2011 at Children's Healthcare of Atlanta.
Groups:
- Rituximab Arm: 375 mg/m2/dose on days 8, 15, 22, and 29 diluted in NS to a final concentration of 1 mg/ml for ease of administration. Administer intravenously through a dedicated line.
Period: Overall Study
Arm/Group | Rituximab Arm
Started | 1
Completed | 0
Not Completed | 1
Not completed — Prescribed exclusion drug | 1

BASELINE CHARACTERISTICS:
Population: no patients were analyzed due to early termination of study
Arm/Group | Rituximab Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: 4 Month Event Free Survival (EFS)
Description: To estimate the 4 month EFS after therapy with rituximab and cytotoxic chemotherapy (prednisone/etoposide/ifosfamide) in patients with second relapse/refractory ALL.
Time Frame: one year after enrollment
Population: The one subject was enrolled became a screen failure as she started a prohibited medication prior to going on study.
Arm/Group | Rituximab Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Toxicities of Rituximab
Description: To describe the toxicities of rituximab in addition to prednisone, etoposide, and ifosfamide.
Time Frame: two months after treatment
Population: The one subject was enrolled became a screen failure as she started a prohibited medication prior to going on study.
Arm/Group | Rituximab Arm
Number analyzed (Participants) | 0

3. Primary Outcome: Remission Induction Rate
Description: To estimate the remission induction rate of the addition of rituximab to cytotoxic chemotherapy (prednisone/etoposide/ifosfamide) in patients with second relapse/refractory ALL.
Time Frame: one month
Population: The one subject was enrolled became a screen failure as she started a prohibited medication prior to going on study.
Arm/Group | Rituximab Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Minimal Residual Disease
Description: To perform serial minimal residual disease (MRD) measurements to provide an objective determination of the effectiveness of this therapy.
Time Frame: one month after treatment
Population: The one subject was enrolled became a screen failure as she started a prohibited medication prior to going on study.
Arm/Group | Rituximab Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Prednisone Effect
Description: To correlate the effect of prednisone on CD20 expression using serial measurements of CD20 expression in leukemic blasts.
Time Frame: one month after treatment
Arm/Group | Rituximab Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The one subject was enrolled became a screen failure as she started a prohibited medication prior to going on study, therefore no serious and other [non-serious] adverse events were collected or assessed as part of the study.
Arm/Group | Rituximab Arm
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The one subject was enrolled became a screen failure as she started a prohibited medication prior to going on study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No